CLINICAL TRIAL: NCT06606899
Title: A Comparative Study Between Efficacy of Combined Oral Melatonin With Nasal Sevoflurane Versus Combined Oral Chloral Hydrate With Nasal Sevoflurane in Sedation of Pre-school Children Undergoing Brain Magnetic Resonance Imaging
Brief Title: A Comparison Between Oral Melatonin With Nasal Sevoflurane Versus Oral Chloral Hydrate With Nasal Sevoflurane in Sedation of Children Undergoing Brain MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, riham fathy galal, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FAMSU R202/2024
Record Dates: First submitted 2024-09-14; First posted 2024-09-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Sedation for Children Undergoing MRI
MeSH Terms: interventions — Melatonin; Chloral Hydrate; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Melatonin (Experimental): Group A: will receive oral Melatonin and nasal Sevoflurane.
  Interventions: Drug: Melatonin 3 MG; Drug: Sevoflurane
- Group Chloral-Hydrate (Experimental): Group B: will receive oral Chloral Hydrate and nasal Sevoflurane.
  Interventions: Drug: Chloral Hydrate; Drug: Sevoflurane

INTERVENTIONS:
Drug: Melatonin 3 MG — Oral syrup melatonin 3 mg
  Other Names: Melatonin
  Arms: Group Melatonin
Drug: Chloral Hydrate — Oral chloral hydrate (50 mg/kg, maximum 2 g)
  Other Names: Cloral hydrate
  Arms: Group Chloral-Hydrate
Drug: Sevoflurane — Inhalational Sevoflurane

SUMMARY:
The patients will be randomized into 2 equal groups by a computer-generated random numbers table, named group A, B.

Group A: will receive oral Melatonin and nasal Sevoflurane. Group B: will receive oral Chloral Hydrate and nasal Sevoflurane. In group A, Approximately 45 to 60 min prior to the intended scan time, the children will be given syrup melatonin 3 mg. Before starting the MRI scan, nasal sevoflurane will be started after positioning of the child at a concentration of 1%.

In Group B, the child will receive oral chloral hydrate (50 mg/kg, maximum 2 g) in syrup form was given to patients requiring sedation. Before starting the MRI scan, nasal sevoflurane will be started after positioning of the child at a concentration of 1% and will be increased gradually as needed to achieve adequate level of sedation.

The child will wait on a general hospital bed in a darkened room with its parents/carers at the rest room. When the radiology technicians decide; the child could be scanned, the child will then be transported in the arms of the parents/carers. Prior to entering the scanning room, the children and parents/carers will be checked for metal to ensure safe entrance. The child will then be lifted from the bed onto the MRI scanning table. Children will be scanned with headphones. If children did not fall asleep or if they woke up.

The MRI scan will be started. After the scanning procedure, the child and its parents/carers will be allowed to go home if the child feels well. All scans will be done on a 1.5 Tesla MR system, using a regular head coil. The MRI studies will be performed during daytime, the protocol duration will range from approximately 10 to 30 min, including positioning of the patient on the scan table. In case children move, radiology technicians could pause the study till the patients is adequately sedated and stops movement. An MRI scan will be considered to have failed when; the entire MRI scan was not assessable because of movement or in the presence of moved scans

DETAILED DESCRIPTION:
The patients will be randomized into 2 equal groups by a computer-generated random numbers table, named group A, B.

Group A: will receive oral Melatonin and nasal Sevoflurane. Group B: will receive oral Chloral Hydrate and nasal Sevoflurane. In group A, Approximately 45 to 60 min prior to the intended scan time, the children will be given syrup melatonin 3 mg. Before starting the MRI scan, nasal sevoflurane will be started after positioning of the child at a concentration of 1%.

In Group B, the child will receive oral chloral hydrate (50 mg/kg, maximum 2 g) in syrup form was given to patients requiring sedation. Before starting the MRI scan, nasal sevoflurane will be started after positioning of the child at a concentration of 1% and will be increased gradually as needed to achieve adequate level of sedation.

The child will wait on a general hospital bed in a darkened room with its parents/carers at the rest room. When the radiology technicians decide; the child could be scanned, the child will then be transported in the arms of the parents/carers. Prior to entering the scanning room, the children and parents/carers will be checked for metal to ensure safe entrance. The child will then be lifted from the bed onto the MRI scanning table. Children will be scanned with headphones. If children did not fall asleep or if they woke up.

The MRI scan will be started. After the scanning procedure, the child and its parents/carers will be allowed to go home if the child feels well. All scans will be done on a 1.5 Tesla MR system, using a regular head coil. The MRI studies will be performed during daytime, the protocol duration will range from approximately 10 to 30 min, including positioning of the patient on the scan table. In case children move, radiology technicians could pause the study till the patients is adequately sedated and stops movement. An MRI scan will be considered to have failed when; the entire MRI scan was not assessable because of movement or in the presence of moved scans

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of anesthesiologists' physical status (ASA) I to II.
2. Aged 2 to 5 years.
3. Both sexes.
4. Patients scheduled for Brain MRI.

Exclusion Criteria:

1. Parent refusal.
2. ASA physical status III or more.
3. Patients with known allergy to any of the study drugs.
4. Children with COSA.
5. Patients with history of cardiovascular disease.
6. Patients older than 5 years.
7. Patients with neuromuscular disease.
8. Patients younger than 2 years.
9. Patients suffering from respiratory tract infection.
10. Patients with family history of malignant hyperthermia.
11. Patients with any Musculoskeletal disorder.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Ramsey sedation scale recorded before starting the MRI exam.Ramsey sedation scale is a 6-point scoring system used to assess a patient's level of arousal and sedation. The scores range from 1 (anxious and agitated) to 6 (unresponsive to pain). | 3 months
  Ramsey sedation scale recorded before starting the MRI exam.
  After completion of data collection, we also analyzed 'Ramsey seadtion scale' because it was clinically relevant but not prospectively specified. This analysis is therefore post-hoc.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided